CLINICAL TRIAL: NCT07326852
Title: Effect of Hybrid Assistive Limb (HAL) Application on Locomotor Function and Balance Parameters in Multiple Sclerosis Patients
Brief Title: Hybrid Assistive Limb Application in Multiple Sclerosis Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mehmet Ozkeskin, Associate Professor of Physical Therapy and Rehabilitation, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOzkeskin25
Record Dates: First submitted 2025-11-18; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; exoskeleton
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MS (Experimental): Participants will receive walking rehabilitation with a lower extremity type Hybrid Assistive Limb (HAL) device, 5 days a week, 1 hour per day, for a total of 2 months.
  Interventions: Device: Hybrid Assistive Limb (HAL)

INTERVENTIONS:
Device: Hybrid Assistive Limb (HAL) — Participants will receive walking rehabilitation with a lower extremity type Hybrid Assistive Limb (HAL) device, 5 days a week, 1 hour per day, for a total of 2 months.

SUMMARY:
The Hybrid Assistive Limb (HAL) exoskeleton detects bioelectrical signals from the muscles, responds to the intention of voluntary movement, and provides biological feedback. In this study, the effects of HAL application on walking performance and balance in patients with multiple sclerosis will be examined in a single-center, controlled design. Participants will undergo walking rehabilitation with HAL for 1 hour per day, 5 days a week, for a total of 2 months. Walking and balance performance will be assessed before and after the intervention using the 10-Minute Walk Test (10MWT) to measure maximum walking speed, the 6-Minute Walk Test (6MWT) to evaluate walking endurance and cardiorespiratory performance, and the Timed Up and Go Test (TUG) to assess functional mobility and dynamic balance. Additionally, walking parameters and static balance will be measured using Tecnobody systems. Appropriate statistical tests will be applied, and a significance level of p<0.05 will be considered.

DETAILED DESCRIPTION:
The Hybrid Assistive Limb (HAL) exoskeleton is a robotic device that detects bioelectrical signals from the muscles, responds to the user's intention to move voluntarily, and provides biological feedback to support motor function. This study aims to investigate the effects of HAL-assisted walking rehabilitation on walking performance and balance in patients with MS in a single-center, controlled design.

Participants will undergo HAL-assisted walking rehabilitation for 1 hour per day, 5 days a week, over a period of 2 months. Assessments will be conducted before and after the intervention by trained clinicians and physiotherapists under standardized conditions. Walking and balance performance will be evaluated using the 10-Minute Walk Test (10MWT) to measure maximum walking speed, the 6-Minute Walk Test (6MWT) to assess walking endurance and cardiorespiratory performance, and the Timed Up and Go Test (TUG) to evaluate functional mobility and dynamic balance. Additionally, walking parameters-including step length, cadence, walking speed, joint range of motion of the hip, knee, and trunk, and gait symmetry-will be analyzed using the Tecnobody Walker View system, while static balance will be measured with the Tecnobody D-Wall system under eyes-open and eyes-closed conditions.

ELIGIBILITY:
Inclusion Criteria:

* No previous robotic rehabilitation.
* Completion of the 10-meter walk test.
* Mini mental status score ≥24.
* MASS score <2.
* EDSS <6.

Exclusion Criteria:

* History of serious degenerative disease.
* Presence of open wounds.
* History of thoracic surgery.
* Chronic respiratory diseases.
* Presence of unstable cardiovascular disease.
* Medical conditions that prevent mobilization.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
10-Meter Walk Test (10mWT) | Baseline (study start) and at 2 months.
  10-Meter Walk Test (10mWT): In this study, the 10-Meter Walk Test (10mWT) will be administered to assess walking speed. Participants will be asked to walk at a comfortable pace along the middle 10-meter section of a 14-meter walkway on level ground.
Timed Up and Go Test (TUG) | Baseline (study start) and at 2 months.
  During the test, participants will be asked to rise from a 47 cm high chair with a backrest and armrests, walk a distance of 3 meters, return to the starting point by turning at a marked cone, and then sit back down in the chair.
6-Minute Walk Test (6MWT) | Baseline (study start) and at 2 months.
  The test will be performed in a straight 30-meter corridor, following the standard protocol established by the American Thoracic Society.
Balance performance assessed using the TecnoBody D-Wall system | Baseline (study start) and at 2 months.
  Balance performance will be evaluated using the TecnoBody D-Wall device (TecnoBody Srl, Bergamo, Italy). The primary balance outcome will be the stability index score obtained from the system. Higher scores indicate better balance performance.
Stride Length Assessed by TecnoBody Walker View | Baseline and at 2 months
  Stride length measured using the TecnoBody Walker View gait analysis system.
Walking Speed Assessed by TecnoBody Walker View | Baseline and at 2 months
  Walking speed will be measured using the TecnoBody Walker View gait analysis system. Participants will walk at a comfortable pace along the walkway, and the average speed in meters per second will be recorded.
Double Support Time Assessed by TecnoBody Walker View | Baseline and at 2 months
  Double support time, defined as the duration when both feet are in contact with the ground during gait, will be measured in seconds using the TecnoBody Walker View system.
Gait Symmetry Index Assessed by TecnoBody Walker View | Baseline and at 2 months
  Gait symmetry will be assessed using the TecnoBody Walker View system by calculating the symmetry index from step length and stance duration for both legs, expressed as a percentage.

SECONDARY OUTCOMES:
Disease severity assessed by the Expanded Disability Status Scale (EDSS) | Baseline (study start) and at 2 months.
  Disease severity will be assessed using the Expanded Disability Status Scale (EDSS), a standardized and validated scale for patients with multiple sclerosis. The EDSS score ranges from 0 to 10, with higher scores indicating greater disability and worse clinical status.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Karşıyaka, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Undecided